CLINICAL TRIAL: NCT03539614
Title: Noradrenergic Biomarkers in PTSD: Precision Medicine & Mechanisms
Brief Title: Predicting Responses to PTSD Treatment With Iris and Cardiovascular Tests
Acronym: PREDICT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MHBB-003-17F; 1IK2CX001774-01 (NIH)
Record Dates: First submitted 2018-05-02; First posted 2018-05-29 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Prazosin; Nightmares; N-of-1
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Prazosin

STUDY DESIGN:
Intervention Model Description: This study is a modified cross-over study, also called an aggregated N-of-1 study. Each participant who meets criteria for participation in and completes the treatment portion of the study will spend time on open-label prazosin, blinded prazosin, and placebo.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: During the portion of the study where participants are receiving either placebo or blinded prazosin, the participants, care providers, and outcomes assessors will all be blinded as to whether the participant is at that time receiving prazosin or placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open label, blinded discontinuation, prazosin, placebo (Experimental): All participants in this study will begin with 8 weeks of active treatment (prazosin), followed by a 4 week "blinded discontinuation" block where they will take a capsule that will start out as active treatment (prazosin), but will at some point change to placebo. Following these phases of the study, participants will be randomized to two arms. In this first arm, participants will spend 4 weeks on active treatment (prazosin), followed by 4 weeks on placebo.
  Interventions: Drug: Prazosin; Drug: Placebo
- Open label, blinded discontinuation, placebo, prazosin (Experimental): All participants in this study will begin with 8 weeks of active treatment (prazosin), followed by a 4 week "blinded discontinuation" block where they will take a capsule that will start out as active treatment (prazosin), but will at some point change to placebo. Following these phases of the study, participants will be randomized to two arms. In this second arm, participants will spend 4 weeks on placebo, followed by 4 weeks on active treatment (prazosin).
  Interventions: Drug: Prazosin; Drug: Placebo

INTERVENTIONS:
Drug: Prazosin — This is an antagonist of the alpha1 receptor for noradrenaline. It is FDA approved for the treatment of hypertension, and has also been used for benign prostatic hypertrophy (BPH). Most recently, it has been found to be helpful for symptoms of PTSD in some but not all participants.
  Other Names: Minipress
Drug: Placebo — This is a capsule containing an inert substance, in order to provide blinding to participants and study staff of when participants are on active medication and when they are not during the later portions of the trial.

SUMMARY:
Posttraumatic stress disorder (PTSD) affects many individuals who experience a traumatic event. There are a variety of treatment options for PTSD, including psychotherapy (talk therapy) options, as well as medications, such as the drug prazosin. Each of the treatment options available is effective at significantly reducing the symptoms of PTSD in some, but not all, individuals with PTSD. However, investigators are not yet able to predict in advance who is likely to respond to which of the available treatments. Neither are the investigators able to explain what changes in the brain after exposure to a traumatic stressors, and why it results in persistent symptoms of PTSD for some people, but not for others.

In this study, the investigators are testing two things: First, is testing whether two simple, easy tests of how an individual's blood pressure changes with standing and how an individual's eye reacts to a pulse of light may be able to predict whether that person is likely to respond to the medication prazosin for PTSD. Second, is testing whether those who have been exposed to a traumatic stress show differences in how their body regulates the response to the stress-signal noradrenaline.

DETAILED DESCRIPTION:
In this study, individuals will undergo an assessment that includes taking a history of their previous exposure to traumatic events, an assessment of current mental health symptoms including those associated with PTSD, and an assessment of physiologic measures, such as blood pressure and pupillary responses to light. For individuals who have current symptoms of PTSD and for whom use of the medication prazosin is a reasonable and safe option, a second phase of the study will be offered. In this second phase, how the individual's PTSD symptoms change when taking prazosin will be assessed. In addition, to test whether any changes are related to the prazosin itself or are part of a placebo effect, the individual will be randomly assigned to periods where he or she is taking a pill that looks like prazosin but is actual placebo (a pill with no active ingredient), and periods where he or she is taking a pill that looks the same but this time is actual prazosin.

Of note, there is also an additional observational portion of the protocol that is not a direct part of the interventional trial described here, but data from which will be used to help to interpret the data from the interventional trial; because reporting of study results depends on both portiosn, the study completion date estimates/reports will reflect when both the interventional and observational trial components are complete.

ELIGIBILITY:
Inclusion Criteria:

* Veteran of the U.S. Armed Forces
* Current diagnosis of PTSD (as documented in clinical chart and/or per participant report; a rule out diagnosis from a VA provider accompanied by a referral to the VA PTSD Outpatient Clinic (POC) will also be considered sufficient for inclusion)
* Woman of childbearing potential must agree to abstain from sexual relations that could result in pregnancy or use an effective method of birth control acceptable to both participant and study clinician during the study. Men are not required to use contraception during the study.

Exclusion Criteria:

* Psychiatric:

  * Any known diagnosis of a primary psychotic or major neurocognitive disorder, including schizophrenia, brief psychotic disorder, or Alzheimer's or other dementia, as well as bipolar type I
  * Severe psychiatric instability or severe situational life crises, including evidence of being actively suicidal or homicidal, or any behavior which poses an immediate danger to participant or others.

    * Note: Nonsuicidal depression comorbid with PTSD will not be exclusionary. Participants may continue in any concurrent psychotherapy or pharmacotherapy in which they are participating, other than pharmacotherapeutic agents specifically listed above. Participants with active suicidal ideation or with depression severe enough to require psychiatric hospitalization will be excluded.
* Medical:

  * Significant bilateral visual loss (would preclude performing the PLR measurements)
  * Current pregnancy or lactation
  * Allergy or previous adverse reaction to prazosin or other alpha-1 antagonist
  * Acute or unstable chronic medical illness, including unstable angina, recent myocardial infarction (within 6 months), congestive heart failure, preexisting hypotension (systolic <110) or orthostatic hypotension (systolic drop > 20mmHg after two minutes standing or any drop accompanied by dizziness); autoimmune disorders; insulin-dependent diabetes
  * Chronic renal or hepatic failure, acute pancreatitis, Meniere's disease, benign positional vertigo, or narcolepsy
* Medication / treatment:

  * Any use within the 7 days prior to baseline of prazosin, doxazosin, clonidine, guanfacine, trazodone, or nonbenzodiazepine hypnotics, and/or unwillingness to avoid these medications for the duration of the study
  * Use of avanafil (Stendra), sildenafil (Viagra), tadalafil (Cialis), and vardenafil (Levitra) will be not be permitted during the study dose titration period because of increased risk of hypotension in combination with alpha-1 blockers, but will be allowed at 1/2 the usual starting dose following dose titration
  * Current use of nitrates, or of alternative medications or supplements with significant vasodilatory properties (e.g., nitrate containing supplements) Participants may also be excluded at the discretion of PI or study clinicians if they appear to be unsuitable for this research study for a reason not detailed here.

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in total PTSD Checklist for DSM 5 (PCL5) score | The PCL5 total score is assessed at baseline, during each stage of the study, and at the endpoint of the study. Thus, measurements will be scheduled to occur at the following time points, relative to the baseline visit: 0, 4, 8, 9-12, 16, and 20 weeks
  The PTSD Checklist for DSM 5 is a self-reported rating scale where an individual rates the severity of each symptom of PTSD on a likert scale. The ratings on individual items are summed to create a total score, which ranges from 0 to 80, with higher scores indicating more symptoms. The relationship between changes in participants' total PCL scores at different time points and prazosin exposure - and whether this relationship is moderated by baseline biomarker values - will be analyzed using a linear mixed effects model.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca C. Hendrickson, MD PhD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No